CLINICAL TRIAL: NCT03973164
Title: Bone Marrow Cytology, Pathology and 18F-FDG PET/CT and Pelvic MRI in the Diagnosis of Lymphoma Bone Marrow Invasion
Brief Title: The Value of Pelvic Magnetic Resonance Imaging in Detecting Bone Marrow Infiltration of Lymphoma
Acronym: PMRIL
Status: Completed | Type: Observational
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Liao, Principal Investigator, Guangxi Medical University
Other Study IDs: Pelvic MRI/lymphoma
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis of lymphoma bone marrow infiltration is very important for the staging and treatment mode of lymphoma. Traditional bone marrow cytology and pathology examinations are only performed locally, and missed diagnosis is possible. The study explore the value of multi-parameter pelvic magnetic resonance in detecting bone marrow infiltration with newly diagnosed lymphoma patients . This study also explore the consistency of pelvic magnetic resonance and PET/CT for detection of lymphoma bone marrow infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Lymphoma subtypes were diagnosed on the basis of tissue samples obtained by biopsy or surgery according to the criteria outlined in the current World Health Organization (WHO) classification of hematologic and lymphoid malignancies, by are reference pathologist.
* Patients who gave written informed consent were referred for MRI.
* Stable physical medical conditions (patients conscious and comfortable, scheduled for an elective diagnostic imaging).

Exclusion Criteria:

• Pregnancy, general contraindications to MRI.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was an Asian race with lymphoma.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Agreement Between MRI and Bone marrow cytology, pathology and follow-up at Diagnosis | Within 30 days prior to start of chemotherapy
  MRI-positive lesions that cannot be confirmed by bone marrow cytology and pathology will be confirmed by MRI follow-up.

SECONDARY OUTCOMES:
Agreement Between MRI and 18F-FDG PET/CT at Diagnosis | Within 30 days prior to start of chemotherapy
  Region based agreement (%; kappa value) of MRI with 18F-FDG PET/CT at diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Tumor Hospital，Guangxi Medical University, Nanning, China

REFERENCES:
- [Background] Barrington SF, Mikhaeel NG, Kostakoglu L, Meignan M, Hutchings M, Mueller SP, Schwartz LH, Zucca E, Fisher RI, Trotman J, Hoekstra OS, Hicks RJ, O'Doherty MJ, Hustinx R, Biggi A, Cheson BD. Role of imaging in the staging and response assessment of lymphoma: consensus of the International Conference on Malignant Lymphomas Imaging Working Group. J Clin Oncol. 2014 Sep 20;32(27):3048-58. doi: 10.1200/JCO.2013.53.5229. PMID 25113771